CLINICAL TRIAL: NCT04603885
Title: Feasibility Testing a Randomized Controlled Trial of an mHealth-enhanced Exercise Program to Improve Cognition for T2DM Patients
Brief Title: Using Polar Unite Fitness Watch to Improve Cognition for T2DM Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Arkansas, Fayetteville (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2009284124
Record Dates: First submitted 2020-10-21; First posted 2020-10-27 (Actual); Last update posted 2020-10-27 (Actual); Status verified 2020-10

CONDITIONS: Diabetes Mellitus, Type 2, Cognitive Dysfunction, Epigenetics, Exercise
MeSH Terms: conditions — Diabetes Mellitus; Cognitive Dysfunction; Motor Activity | interventions — Muscle Stretching Exercises

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aerobic exercise group (Experimental): Aerobic exercise will be measured with a Polar United fitness watch. Heart rate during exercise will be measured using a Polar United fitness watch, which has been validated for monitoring moderate and high intensity physical activity.
  Interventions: Behavioral: Aerobic exercise program
- Attention control group (Placebo Comparator): The time-equivalent, stretching movements will serve as the placebo exercise condition in this proposed study. Previous research has shown that stretching could reduce attrition and patient dissatisfaction and better ensure allocation concealment. Following baseline measures, a student will demonstrate the use of a Polar United fitness watch and stretching movements via zoom from week 3 to week 5. Starting on week 3, participants will perform the prescribed stretching exercise 3 times a week, maintaining heart rate below 40% of heart rate reserve during exercise.
  Interventions: Behavioral: Stretching exercise

INTERVENTIONS:
Behavioral: Aerobic exercise program — A randomized controlled trial will be used to test the feasibility of a home-based exercise program to improve BDNF DNA demethylation among individuals with T2DM. A total of 42 participants will be randomized 2:1 to receive aerobic exercise intervention (n=28) or attention control (n=14) for 3 months. This ratio is used to offset an anticipated attrition imbalance across groups.
  Arms: Aerobic exercise group
Behavioral: Stretching exercise — stretching exercise
  Arms: Attention control group

SUMMARY:
Type 2 diabetes mellitus (T2DM) impairs the brain, leading to cognitive dysfunction, which carries substantial lifetime consequences. This highlights an urgent need to find effective therapeutic strategies to improve cognitive function among those with T2DM. Aerobic exercise enhances cognitive function among healthy subjects through increased release of BDNF. BDNF supports survival of existing neurons and promotes growth of new neurons and synapses. Emerging evidence suggests that reduced BDNF levels may exacerbate cognitive dysfunction associated with T2DM. Compared to drug delivery of BDNF, aerobic exercise is a low-cost, safe, and easily accessible path to increasing endogenous BDNF levels. One critical genetic variant that affects BDNF secretion and cognition is the BDNF Val66Met variant, which is a common missense polymorphism that results in a valine (Val) to methionine (Met) substitution at codon 66 located in exon IX of the BDNF gene. The Met allele alters intracellular processing, trafficking, packaging of pro-BDNF, and consequently interferes with the activity-dependent secretion of mature BDNF among Met carriers. In addition, previous research reported an influence of the Val66Met variant on the methylation level of the surrounding region. Carrying a G nucleotide (i.e., Val allele) will have an additional CpG site, and Val/Val homozygotes demonstrated a significant increase in methylation levels of four nearby CpG sites compared to Val/Met heterozygotes and Met/Met homozygotes. Because high BDNF gene methylation is associated with reduced BDNF mRNA levels, this may result in lower BDNF levels among Val/Val carriers. However, the transcription of promoter IV can be initiated by exercise, suggesting that epigenetic modulation of BDNF gene expression may be achieved by exercise. It is plausible that exercise may partly reverse transcriptional repression through dynamic DNA demethylation, but the interaction between DNA demethylation and Val homozygosity may be different from that in Met/Met and in Val/Met carriers, which could explain interpersonal differences in cognitive outcomes among these carriers following exercise training. So far, the evidence on the interplay of the Val66Met polymorphism, DNA methylation, and exercise on cognition among individuals with T2DM is still lacking. A total of 42 participants with T2DM will be randomized 2:1 to receive aerobic exercise intervention (n=28) or attention control (n=14) for 3 months. Both groups will receive weekly phone calls during the intervention and standard printed education materials regarding diabetes self-management. In addition to these interventions, the aerobic exercise group (i.e., experimental group) will also perform home-based walking exercise, while the attention control group will perform home-based stretching exercise. Trained students will monitor the exercise sessions for both groups at the Connected Health Platform (hereafter referred to as "platform"). Blood samples will be collected at baseline and three months. Outcomes of interest include post-intervention changes in plasma BDNF levels, BDNF DNA methylation executive function, memory, and processing speed. The study will evaluate the feasibility of the home-based exercise intervention. The study will also evaluate preliminary effectiveness of the supervised exercise program on of the exercise program on BDNF DNA demethylation. An exploratory aim is to explore the association of DNA demethylation with plasma BDNF levels and cognition.

ELIGIBILITY:
Inclusion Criteria:

* Participants eligible for this study will be physically inactive adults with no major chronic physical or mental disorders but classified as having low physical activity levels determined by the International Physical Activity Questionnaire. Participants must have a documented medical diagnosis of T2DM and must be receiving diabetes care at the time of enrollment. Participants must be English-speaking and are able to give informed consent.

Exclusion Criteria:

* Exclusion criteria include uncontrolled hypertension with resting blood pressure of 160/90 mmHg or higher, having symptoms of coronary ischemia such as chest pain and severe shortness of breath during activities of daily living, loss of consciousness/fainting for any reason, or having any other medical or physical conditions that may interfere with exercise participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2020-10-27 (Estimated); Primary Completion 2021-05-15 (Estimated); Study Completion 2021-07-15 (Estimated)

PRIMARY OUTCOMES:
BDNF DNA demethylation in percentage | Three months

SECONDARY OUTCOMES:
Plasma BDNF levels in ng | Three months
Executive function | Three months
  Executive function will be measured by the Dimensional Change Card Sort Test. Test-retest reliability of the test is 0.88. Convergent validity and discriminant validity is -0.51 and 0.14, respectively.
Episodic memory | Three months
  Episodic memory will be measured by the Picture Sequence Memory Test. Test-retest reliability of the test is 0.77. Convergent validity and discriminant validity is 0.69 and -0.08, respectively.
Working memory | Three months
  Working memory will be measured by the List Sorting Working Memory Test. Test-retest reliability of the test is 0.77. Convergent validity and discriminant validity are 0.58 and 0.30, respectively.
Processing speed | Three months
  Processing speed will be measured by the Pattern Comparison Processing Speed Test. The test takes about 3 minutes to compete. Test-retest reliability of the test is 0.72. Convergent validity and discriminant validity is 0.49 and 0.12, respectively.

IPD SHARING:
Plan to Share IPD: No